CLINICAL TRIAL: NCT03972670
Title: Correlation Between Postoperative Central Corneal Thickness and Endothelial Damage After Cataract Surgery by Phacoemulsification
Brief Title: Correlation Between Postoperative Central Corneal Thickness and Endothelial Damage After Cataract Surgery
Acronym: ECOCHI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-13Obs-CHRMT
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Cataract; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study correlation between postoperative corneal edema and endothelial cell loss after cataract surgery by microcoaxial phacoemulsification.

DETAILED DESCRIPTION:
Cataract surgery facilitates improved visual acuity through extraction of an opacified lens, followed by intraocular lens implantation. An average adult cornea has 2000 to 2500 cells/mm2, a count that diminishes with age with a rate of attrition of approximately 0.3% to 0.5% per year. Long-term postoperative corneal transparency depends on the morphological stability and functional integrity of the corneal endothelium. It is well established that all surgical interventions that require entry into the anterior chamber result in some damage to the corneal endothelium.

Endothelial cell loss results in cell hypertrophy to maintain continuity, resulting in a change in endothelium cell density and morphology. Many studies have assessed the impact of various surgical techniques on endothelial damage and numerous studies have investigated the factors influencing endothelial cell loss after phacoemulsification. The goal of this study is to investigate the correlation of postoperative corneal edema with the reduction of endothelial corneal cell density after phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* The presence of senile cataract with equivalent grades and a history of visual acuity regression

Exclusion Criteria:

* Patient with total white cataract
* With history of ocular surgery
* With other eye diseases (corneal pathology, Fuchs dystrophy, uveitis and glaucoma) or systemic diseases (diabetic disorder and dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery were older than 18 years. Subjects had cataract up to C5, N4 and P5 on the LOCS III classification
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Pachymetry | Day 1
  Measurement of the thickness of the eye's cornea with a pachymeter

SECONDARY OUTCOMES:
Endothelial cell density | Day 1
  Endothelial cell density measurements with noncontact specular microscope
Pachymetry after 1 month | Day 30
  Measurement of the thickness of the eye's cornea with a pachymeter
Endothelial cell density after 1 month | Day 30
  Endothelial cell density measurements with noncontact specular microscope